CLINICAL TRIAL: NCT04638361
Title: Prevalence of Laryngeal Disorders After Childhood Cardiac Surgery and Evaluation of Their Long-term Recovery
Brief Title: Laryngeal Disorders After Childhood Cardiac Surgery
Acronym: RECUP-TML
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0505; 2020-A01701-38 (Other: ID-RCB)
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Laryngeal Injury; Swallowing Disorder; Voice Disorders in Children; Surgery--Complications
Keywords: Laryngeal dysfunction; Cardiac surgery
MeSH Terms: conditions — Deglutition Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No laryngeal mobility disorder post cardiac surgery: No Follow up, no questionnaires and no nasofibroscopic control.
- Laryngeal mobility disorder post cardiac surgery: During a follow-up consultation, questionnaires will be offered to assess the child's quality of life.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — To explore the quality of life, two questionnaires will be submitted to the parents and the child. The first one is the pediatric version of the VHI (Voice Handicap Index), which explore, using 23 items, the functional, physical and emotional aspects of the dysphonia. The second one is the PEDI-EAT-10 (Pediatric Voice Handicap Index - Eating Assessment Tool), which explore, through 10 items (ranging from 0 to 4), the risk of aspiration and assess the impact of possible dysphagia on quality of life.
  Groups: Laryngeal mobility disorder post cardiac surgery

SUMMARY:
Laryngeal disorders after childhood cardiac surgery is a complication well described in the literature. However, the long term progression of the affected children has never been studied (all the studies stopped before 2 years of follow up).

ELIGIBILITY:
Inclusion Criteria:

* No opposition from children and parents
* Patient or parents able to understand the ins and outs of the study

Exclusion Criteria:

* None

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 5 and 10 years old, having undergone a nasofibroscopy following cardiac surgery performed before their first year of life (between 01/01/2010 and 12/31/2015).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Prevalence of a laryngeal mobility disorder after childhood cardiac surgery | One day
  The prevalence will be evaluated on the respiratory, food or phonatory difficulties reported after surgery as well as on the result of early postoperative nasofibroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia AYARI-KHALFALLAH, MD, Principal Investigator — Hôpital Femme Mère Enfant - Department of ENT Pediatric surgery,
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France